CLINICAL TRIAL: NCT01774955
Title: The GReek AntiPlatElet (GRAPE) Registry: A Multicenter Observational Prospective Investigation of Antiplatelet Treatment in Patients With Acute Coronary Syndrome Subjected to Percutaneous Coronary Intervention
Acronym: GRAPE
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Collaborators: Hellenic Cardiology Society (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, University of Patras
Other Study IDs: GRAPE registry
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicenter, prospective, observational investigation, focusing of antiplatelet treatment in patients with moderate to high risk acute coronary syndrome (TIMI risk score ≥3)subjected to percutaneous coronary intervention (PCI), being conducted in 7 PCI capable hospitals in Greece. Data concerning patients' demographic, clinical/procedural characteristics and contraindications/special warnings and precautions to P2Y12 inhibitors are collected during initial hospitalization. Study involves 3 follow-up visits after hospital discharge(Day 30, at 6 months and at 12 months) where data on major adverse cardiac events (death, myocardial infarction, stroke, urgent revascularization procedure with PCI or CABG), bleeding events(according to Bleeding Academic Research Consortium criteria)and adherence to antiplatelet treatment are collected.

In patients under ticagrelor or prasugrel treatment, platelet reactivity measurement with VerifyNow assay will be performed at Day 30

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Acute coronary syndrome moderate to high risk (TIMI risk score ≥3) subjected to PCI
* Informed consent

Exclusion Criteria:

* Pregnancy/Breastfeeding
* Inability to give informed consent
* High probability of being unavailable for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is consisted of patients with acute coronary syndrome subjected to PCI in 6 geographic regions of Greece
Sampling Method: Probability Sample
Enrollment: 2047 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MACES at 12 months following PCI | 12 months
  The composite of death, myocardial infarction, stroke, urgent revascularization procedure with PCI or CABG at 12 months after PCI

SECONDARY OUTCOMES:
Any bleeding event (BARC classification) at 12 months after PCI | 12 months
  Any bleeding event (BARC classification) at 12 months after PCI

OTHER OUTCOMES:
Rates of P2Y12 inhibitors (Clopidogrel, Prasugrel and Ticagrelor) use at 12 months following PCI | 12 months
  Rates of P2Y12 inhibitors (Clopidogrel, Prasugrel and Ticagrelor) use at 12 months following PCI
Any bleeding event (BARC classification) at 12 months after PCI | 1 year
  Any bleeding event (BARC classification) at 12 months after PCI between lowest and highest quartile of platelet reactivity value at Day 30

CONTACTS AND LOCATIONS:
Locations (9):
- Greece (9):
  - Patras University Hospital, Pátrai, Achaia
  - G.Gennimatas General Hospital, Athens, Attica
  - University Hospital, Alexandroupolis, Alexandroupoli
  - 1st Department of Cardiology, Ippokration Hospital, Athens
  - Alexandra Hospital, Athens, Greece, Athens
  - Onassis Cardiac Surgery Center, Athens
  - University Hospital, Ioannina, Ioannina
  - Iraklion University Hospital, Iraklion, Greece, Irakleio
  - Larissa University Hospital, Larissa

REFERENCES:
- [Derived] Alexopoulos D, Vogiatzi C, Stavrou K, Vlassopoulou N, Perperis A, Pentara I, Xanthopoulou I. Diabetes mellitus and platelet reactivity in patients under prasugrel or ticagrelor treatment: an observational study. Cardiovasc Diabetol. 2015 May 30;14:68. doi: 10.1186/s12933-015-0232-1. PMID 26025572
- [Derived] Alexopoulos D, Stavrou K, Koniari I, Gkizas V, Perperis A, Kontoprias K, Vogiatzi C, Bampouri T, Xanthopoulou I. Ticagrelor vs prasugrel one-month maintenance therapy: impact on platelet reactivity and bleeding events. Thromb Haemost. 2014 Sep 2;112(3):551-7. doi: 10.1160/TH14-02-0119. Epub 2014 Jul 3. PMID 24990396
- [Derived] Alexopoulos D, Goudevenos JA, Xanthopoulou I, Deftereos S, Sitafidis G, Kanakakis I, Hamilos M, Parissis H, Ntalas IV, Angelidis C, Petousis S, Vavuranakis M, Hahalis G, Stefanadis C; GRAPE Investigators. Implementation of contemporary oral antiplatelet treatment guidelines in patients with acute coronary syndrome undergoing percutaneous coronary intervention: a report from the GReek AntiPlatelet rEgistry (GRAPE). Int J Cardiol. 2013 Oct 15;168(6):5329-35. doi: 10.1016/j.ijcard.2013.08.007. Epub 2013 Aug 15. PMID 23978364